CLINICAL TRIAL: NCT01041378
Title: Efficacy of Intravenous Dexamethasone on Postoperative Caudal Analgesia in Pediatric Orchiopexy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Kil Hae Keum / Professor of Anesthesiology and Pain Medicine at Severance Hospital, Yonsei University Health System
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 4-2009-0558
Record Dates: First submitted 2009-12-30; First posted 2009-12-31 (Estimated); Last update posted 2010-06-16 (Estimated); Status verified 2010-05

CONDITIONS: Pain
Keywords: Pediatric patients (6 months-5 years) scheduled elective day-case orchiopexy
MeSH Terms: conditions — Pain | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: dexamethasone — Intravenous dexamethasone (0.5mg/kg) before incision

SUMMARY:
The purpose of this study is to evaluate postoperative pain control for pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients scheduled for elective day-case orchiopexy.

Exclusion Criteria:

* Infants or children with history of steroid allergy, renal, hepatic disease, or contraindication for caudal analgesia.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2010-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Children's Hospital of Eastern Ontario Pain Scale, CHEOPS and Faces, Legs, Activity, Cry, and Consolability, FLACC | postoperative 24 hours

REFERENCES:
- [Derived] Hong JY, Han SW, Kim WO, Kim EJ, Kil HK. Effect of dexamethasone in combination with caudal analgesia on postoperative pain control in day-case paediatric orchiopexy. Br J Anaesth. 2010 Oct;105(4):506-10. doi: 10.1093/bja/aeq187. Epub 2010 Jul 20. PMID 20659915